CLINICAL TRIAL: NCT00531973
Title: Liposomal Doxorubicin-Investigational Chemotherapy-Tissue Doppler Imaging Evaluation (LITE) Randomized Pilot Study
Brief Title: A Study of Liposomal Doxorubicin in Women With Breast Cancer Exploiting Tissue Doppler Imaging
Acronym: LITE
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Catholic University, Italy (Other)
Collaborators: Cephalon (Industry)
Responsible Party: Marzia Lotrionte, Consultant, Catholic University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: LITE Randomized Pilot Study
Record Dates: First submitted 2007-09-18; First posted 2007-09-19 (Estimated); Last update posted 2009-02-18 (Estimated); Status verified 2009-02

CONDITIONS: Breast Cancer
Keywords: breast cancer; echocardiography; neoplasia
MeSH Terms: conditions — Breast Neoplasms; Neoplasms | interventions — liposomal doxorubicin; Epirubicin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): Liposomal doxorubicin
  Interventions: Drug: liposomal doxorubicin
- B (Active Comparator): epirubicin
  Interventions: Drug: epirubicin

INTERVENTIONS:
Drug: liposomal doxorubicin — 5-fluorouracil (500 mg/m²) + pegylated liposomal doxorubicin (50 mg/m²) + cyclophosphamide (500 mg/m²) + adjuvant radiation therapy ± endocrinological therapy (FalipoC)
  Arms: A
Drug: epirubicin — 5-fluorouracil (500 mg/m²) + epirubicin (90 mg/ m²) + cyclophosphamide (500 mg/ m²) + adjuvant radiation therapy ± endocrinological therapy (FEC90)
  Arms: B

SUMMARY:
The randomized LITE study will compare liposomal doxorubin versus standard epirubicin in the treatment of female breast cancer. In order to detect as early as possible post-chemotherapy cardiotoxicity, tissue Doppler imaging parameters elicited at transthoracic echocardiography will be used and will constitute the primary and co-primary end-points.

DETAILED DESCRIPTION:
The randomized LITE study will compare liposomal doxorubin versus standard epirubicin within a comprehensive adjuvant or neo-adjuvant chemotherapy regimen in women undergoing treatment for breast cancer. The study will enrol a total of 80 patients, randomized 1:1 to liposomal doxorubin vs epirubicin. Standard and tissue Doppler imaging parameters will be appraised at transthoracic echocardiography will be used and will constitute the primary and co-primary end-points. In addition, other efficacy and safety end-points will be appraised, including disease free progression.

ELIGIBILITY:
Inclusion Criteria:

* women with age ≥18 and ≤65 years
* histological and/or cytological diagnosis of clinically non-metastatic breast cancer (c/pTall, c/pNall, cM0)
* indication for integrated treatment with surgical intervention associated with adjuvant or neo-adjuvant chemotherapy, endocrinological and radiation therapy, including adjuvant or neo-adjuvant chemotherapy with anthracycline
* ECOG (Eastern Cooperative Oncology Group) performance status ≤2
* normal kidney, hepatic and hematological function
* normal LV ejection fraction at baseline (≥50%)
* negative pregnancy test in fecund women

Exclusion Criteria:

* metastatic breast cancer
* past radiation therapy and chemotherapy
* hypertension and other cardiovascular risk factors
* prior valvular heart disease
* cardiomyopathy
* chronic or acute congestive heart failure
* LV systolic dysfunction (ejection fraction<50%)
* abnormal complete blood count
* pregnancy
* breast-feeding

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2007-01; Primary Completion 2008-08 (Estimated); Study Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
Comparison of changes of PW-TDI systolic function parameters. The co-primary end-point ill be the comparison of changes from baseline to 12-month follow-up of PW-TDI diastolic function parameters. | Up to 12 months

SECONDARY OUTCOMES:
Changes of standard 2-dimensional echocardiography parameters, including LV ejection fraction, peak values of biochemical markers of cardiac damage and heart failure, ie cardiac troponin T and BNP. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Marzia Lotrionte, MD, Principal Investigator — marzial76@yahoo.it
Locations (1):
- Catholic University, Rome, RM, Italy

REFERENCES:
- [Derived] Lotrionte M, Palazzoni G, Natali R, Comerci G, Abbate A, Di Persio S, Biondi-Zoccai GG. Appraising cardiotoxicity associated with liposomal doxorubicin by means of tissue Doppler echocardiography end-points: rationale and design of the LITE (Liposomal doxorubicin-Investigational chemotherapy-Tissue Doppler imaging Evaluation) randomized pilot study. Int J Cardiol. 2009 Jun 12;135(1):72-7. doi: 10.1016/j.ijcard.2008.03.036. Epub 2008 Jun 24. PMID 18572266